CLINICAL TRIAL: NCT02091622
Title: Increasing the Number of Patients Receiving Information About Transition to End-of-life Care: the Effect of a Half-day Physician and Nurse Training
Brief Title: Increasing the Number of Patients Receiving Information About Transition to End-of-life Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Intervention-sv-pall
Record Dates: First submitted 2014-03-13; First posted 2014-03-19 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Palliative Care; Disclosure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educative intervention (Other): Two municipalities (in charge of nursing homes) and two hospitals were randomized to receive an interactive half-day course about ITEOL for physicians and nurses.
  Interventions: Other: Educative intervention
- No intervention (No Intervention): No intervention.

INTERVENTIONS:
Other: Educative intervention — Two municipalities (in charge of nursing homes) and two hospitals were randomized to receive an interactive half-day course about ITEOL for physicians and nurses.
  Arms: Educative intervention

SUMMARY:
Introduction: Honest prognostication and information for patients are important parts of end-of-life care. This study examined whether an educational intervention could increase the proportion of patients who received information about the transition to end-of-life care (ITEOL).

Method: Two municipalities (in charge of nursing homes) and two hospitals were randomized to receive an interactive half-day course about ITEOL for physicians and nurses. The proportion of patients who received ITEOL was measured with data from the Swedish Register of Palliative Care (SRPC). Patients were only included if they died an expected death and maintained their ability to express their will until days or hours before their death. Four hospitals and four municipalities were assigned controls, matched by hospital size, population, and proportion of patients receiving ITEOL at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Hospitals and municipalities: Participation in the Swedish Register of Palliative Care.
* Patients: Reported from an included hospital or municipality during six months before to six months after intervention.

Exclusion Criteria:

* Hospitals and municipalities: Exclusion criteria were more than 40% patients receiving ITEOL at start of study, too large for an intervention due to practical reasons (university hospitals or municipalities with over 100 000 inhabitants), and hospitals not containing both internal medicine and surgery departments.
* Patients were excluded when death was unexpected, when a forensic post mortem examination was performed, or when the patients had lost their ability to express their will and take part in decisions concerning the content of medical care one week or more before death.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1431 (Actual)
Dates: Start 2011-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who received ITEOL | Six months after intervention
  The proportion of patients who received ITEOL was measured with data from the Swedish Register of Palliative Care (SRPC). Six months after the intervention data were collected from the SRPC for all patients who had died at the included hospitals and municipalities. Data were collected from six months before the intervention to six months after the intervention. The outcome was compared before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Bertil Axelsson, MD PhD, Principal Investigator — Umeå University
Locations (1):
- Umeå University, Dept of radiation sciences, Umeå, Umeå, Sweden